CLINICAL TRIAL: NCT01555151
Title: A Randomized, Double-blind, Double-dummy, 4-week Treatment, Parallel-group Study to Evaluate the Efficacy and Safety of Two Doses of Mometasone Furoate Delivered Via Concept1 or Twisthaler® in Adult and Adolescent Patients With Persistent Asthma
Brief Title: Safety and Efficacy of Mometasone Furoate Delivered Via Concept1 Device or Twisthaler® Device in Adult and Adolescent Patients With Persistent Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CQMF149E2201; 2011-005100-14 (EudraCT Number)
Record Dates: First submitted 2012-03-13; First posted 2012-03-15 (Estimated); Results first posted 2014-08-01 (Estimated); Last update posted 2015-05-01 (Estimated); Status verified 2015-04

CONDITIONS: Asthma
Keywords: Asthma
MeSH Terms: conditions — Asthma | interventions — Mometasone Furoate; QMF149

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Mometasone furoate 80 μg (Experimental): Description: Mometasone furoate (MF) 800 ug delivered via the Twisthaler® device for 2 weeks, followed by MF 200 ug delivered via the Twisthaler® device for 2 weeks or no treatment for 2 weeks, then randomized to MF 80 ug delivered via the Concept1 device for 4 weeks.
  Interventions: Drug: Mometasone furoate; Device: Concept 1
- Mometasone furoate 200 µg (Experimental): Mometasone furoate (MF) 800 ug delivered via the Twisthaler® device for 2 weeks, followed by MF 200 ug delivered via the Twisthaler® device for 2 weeks or no treatment for 2 weeks, then randomized to MF 200 ug delivered via the Twisthaler® device for 4 weeks.
  Interventions: Drug: Mometasone furoate; Device: Twisthaler
- Mometasone furoate 320 µg (Experimental): Mometasone furoate (MF) 800 ug delivered via the Twisthaler® device for 2 weeks, followed by MF 200 ug delivered via the Twisthaler® device for 2 weeks or no treatment for 2 weeks, then randomized to MF 320 ug delivered via the Concept1 device for 4 weeks.
  Interventions: Drug: Mometasone furoate; Device: Concept 1
- Mometasone furoate 800 µg (Experimental): Mometasone furoate (MF) 800 ug delivered via the Twisthaler® device for 2 weeks, followed by MF 200 ug delivered via the Twisthaler® device for 2 weeks or no treatment for 2 weeks, then randomized to MF 800 ug delivered via the Twisthaler® device for 4 weeks.
  Interventions: Drug: Mometasone furoate; Device: Twisthaler

INTERVENTIONS:
Drug: Mometasone furoate — Mometasone furoate (MF) 80 µg once daily delivered via Concept1 device; MF 200 μg once daily delivered via Concept1 device; MF 320μg once daily delivered via Twisthaler® device or 800 μg once daily delivered via Twisthaler® device
  Other Names: QMF149
Device: Concept 1 — A single dose dry powder inhaler (SDDPI)
  Arms: Mometasone furoate 320 µg; Mometasone furoate 80 μg
Device: Twisthaler — A single dose dry powder inhaler (SDDPI)
  Arms: Mometasone furoate 200 µg; Mometasone furoate 800 µg

SUMMARY:
The purpose of this study is to compare the efficacy, safety and pharmacokinetics of Mometasone furoate delivered via Concept1 device or Twisthaler® device in adult and adolescent patients with persistent asthma.

ELIGIBILITY:
Inclusion Criteria:

* Males or females who were ≥ 12 years old at the time informed consent was obtained
* Patients with persistent asthma, diagnosed according to GINA 2010 guideline and who additionally met the following criteria
* Patients who were receiving ICS treatment up to the maximum dose per day as indicated in the corresponding package leaflet and also a stable ICS regimen for at least 4 weeks prior to screening (Visit 2).
* Patients whose level of asthma control according to GINA 2010 guideline was "Partly Controlled" or "Uncontrolled" at screening (Visit 2).
* Patients with a pre-bronchodilator FEV1 value of ≤ 80% of predicted normal value at screening (Visit 2).
* Patients who demonstrated an increase of ≥ 12% and 200 mL in FEV1 over prebronchodilator value within 30 minutes after inhalation of 400 μg of salbutamol (360 μg of albuterol) at Visit 2 or between Visit 2 and Visit 5.
* Patients who were confirmed as "ICS sensitive" by ACQ-5 and FEV1 at Visit 5.

Key exclusion criteria included:

* Patients diagnosed with COPD as defined by the Global Initiative for Chronic Obstructive Lung Disease, updated 2010.
* Patients with concomitant pulmonary disease, pulmonary tuberculosis (unless confirmed by chest X-ray to be no longer active), or clinically significant bronchiectasis.
* Patients with any chronic conditions affecting the respiratory tract (e.g., chronic sinusitis) or chronic lung diseases, which in the opinion of the investigator may interfere with the study evaluation or optimal participation in the study.
* Patients with seasonal allergy which is likely to deteriorate his/her asthma condition during the study period judged by the investigator.
* Patients who have had a severe asthma attack/exacerbation requiring hospitalization in the 6 months prior to Visit 1 or any time between Visit 1 and Visit 5 must discontinue from the trial (screening failure).
* Patients who have had an emergency room visit for an asthma attack/exacerbation within 4 weeks prior to Visit 1 or any time between Visit 1 and Visit 5 must discontinue from the trial (screening failure).
* Patients who have ever required intubation for a severe asthma attack/exacerbation.
* Patients who have had a respiratory tract infection within 6 weeks prior to Visit 1, or any time between Visit 1 and Visit 5 must discontinue from the trial (screening failure).

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 739 (Actual)
Dates: Start 2012-07; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (137):
- Belgium (2):
  - Novartis Investigative Site, Kortrijk, Belgium
  - Novartis Investigative Site, Liège, Belgium
- Canada (6):
  - Novartis Investigative Site, Niagara Falls, Ontario
  - Novartis Investigative Site, Windsor, Ontario
  - Novartis Investigative Site, Mirabel, Quebec
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Québec, Quebec
  - Novartis Investigative Site, Trois-Rivières, Quebec
- Estonia (3):
  - Novartis Investigative Site, Kohtla-Järve, Estonia
  - Novartis Investigative Site, Tallinn, Estonia
  - Novartis Investigative Site, Tartu, Estonia
- Germany (12):
  - Novartis Investigative Site, Berlin, Germany
  - Novartis Investigative Site, Essen, Germany
  - Novartis Investigative Site, Hamburg, Germany
  - Novartis Investigative Site, Leipzig, Germany
  - Novartis Investigative Site, Lübeck, Germany
  - Novartis Investigative Site, Reinfeld, Germany
  - Novartis Investigative Site, Schwerin, Germany
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Goch
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, München
- Hungary (22):
  - Novartis Investigative Site, Balassagyarmat, Hungary
  - Novartis Investigative Site, Budapest, Hungary
  - Novartis Investigative Site, Cegléd, Hungary
  - Novartis Investigative Site, Debrecen, Hungary
  - Novartis Investigative Site, Komárom, Hungary
  - Novartis Investigative Site, Monor, Hungary
  - Novartis Investigative Site, Nyíregyháza, Hungary
  - Novartis Investigative Site, Százhalombatta, Hungary
  - Novartis Investigative Site, Szeged, Hungary
  - Novartis Investigative Site, Szikszó, Hungary
  - Novartis Investigative Site, Törökbálint, Hungary
  - Novartis Investigative Site, Baja
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Gödöllő
  - Novartis Investigative Site, Győr
  - Novartis Investigative Site, Gyula
  - Novartis Investigative Site, Kistelek
  - Novartis Investigative Site, Makó
  - Novartis Investigative Site, Mohács
  - Novartis Investigative Site, Mosonmagyaróvár
  - Novartis Investigative Site, Nagykanizsa
  - Novartis Investigative Site, Szombathely
- India (10):
  - Novartis Investigative Site, Jaipur, India
  - Novartis Investigative Site, Karamsad, India
  - Novartis Investigative Site, Ludhiana, India
  - Novartis Investigative Site, Nagpur, India
  - Novartis Investigative Site, Thrissur, India
  - Novartis Investigative Site, Bangalore, Karnataka
  - Novartis Investigative Site, Mysore, Karnataka
  - Novartis Investigative Site, Pune, Maharashtra
  - Novartis Investigative Site, Coimbatore, Tamil Nadu
  - Novartis Investigative Site, Vellore, Tamil Nadu
- Japan (21):
  - Novartis Investigative Site, Toon-shi, Ehime
  - Novartis Investigative Site, Mizunami, Gifu
  - Novartis Investigative Site, Fukuyama-shi, Hiroshima
  - Novartis Investigative Site, Kitahiroshima-shi, Hokkaido
  - Novartis Investigative Site, Obihiro-shi, Hokkaido
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Tomakomai, Hokkaido
  - Novartis Investigative Site, Kobe, Hyōgo
  - Novartis Investigative Site, Kawasaki-shi, Kanagawa
  - Novartis Investigative Site, Kurashiki, Okayama-ken
  - Novartis Investigative Site, Kurashiki-shi, Okayama-ken
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Sakai, Osaka
  - Novartis Investigative Site, Suita, Osaka
  - Novartis Investigative Site, Toyonaka, Osaka
  - Novartis Investigative Site, Chiyoda-ku, Tokyo
  - Novartis Investigative Site, Chuo-ku, Tokyo
  - Novartis Investigative Site, Hachiōji, Tokyo
  - Novartis Investigative Site, Shinagawa-ku, Tokyo
  - Novartis Investigative Site, Tachikawa, Tokyo
  - Novartis Investigative Site, Toshima-ku, Tokyo
- Latvia (4):
  - Novartis Investigative Site, Rēzekne, LV
  - Novartis Investigative Site, Riga, LV
  - Novartis Investigative Site, Talsi, LV
  - Novartis Investigative Site, Riga
- Lithuania (5):
  - Novartis Investigative Site, Kaunas, LT
  - Novartis Investigative Site, Klaipėda, LT
  - Novartis Investigative Site, Kaunas
  - Novartis Investigative Site, Klaipėda
  - Novartis Investigative Site, Vilnius
- Malaysia (3):
  - Novartis Investigative Site, Kota Kinabalu, Malaysia
  - Novartis Investigative Site, Kuching, Sarawak
  - Novartis Investigative Site, Kuala Lumpur
- Netherlands (7):
  - Novartis Investigative Site, Almere Stad, The Netherlands
  - Novartis Investigative Site, Eindhoven, The Netherlands
  - Novartis Investigative Site, Leiderdorp, The Netherlands
  - Novartis Investigative Site, Rotterdam, The Netherlands
  - Novartis Investigative Site, Zoetermeer, The Netherlands
  - Novartis Investigative Site, Geleen
  - Novartis Investigative Site, Hoofddorp
- Poland (9):
  - Novartis Investigative Site, Bialystok, Poland
  - Novartis Investigative Site, Katowice, Poland
  - Novartis Investigative Site, Krakow, Poland
  - Novartis Investigative Site, Lodz, Poland
  - Novartis Investigative Site, Poznan, Poland
  - Novartis Investigative Site, Warsaw, Poland
  - Novartis Investigative Site, Wroclaw, Poland
  - Novartis Investigative Site, Gdansk
  - Novartis Investigative Site, Skierniewice
- Russia (6):
  - Novartis Investigative Site, Saint Petersburg, Nizhny Novgorod Oblast
  - Novartis Investigative Site, Kazan', Russia
  - Novartis Investigative Site, Moscow, Russia
  - Novartis Investigative Site, Saint Petersburg, Russia
  - Novartis Investigative Site, Yekaterinburg, Russia
  - Novartis Investigative Site, Yaroslavl
- Slovakia (13):
  - Novartis Investigative Site, Bojnice, Slovak Republic
  - Novartis Investigative Site, Bratislava, Slovak Republic
  - Novartis Investigative Site, Košice, Slovak Republic
  - Novartis Investigative Site, Levice, Slovak Republic
  - Novartis Investigative Site, Liptovský Hrádok, Slovak Republic
  - Novartis Investigative Site, Nitra, Slovak Republic
  - Novartis Investigative Site, Rožňava, Slovak Republic
  - Novartis Investigative Site, Šurany, Slovak Republic
  - Novartis Investigative Site, Trenčín, Slovak Republic
  - Novartis Investigative Site, Martin, Slovakia
  - Novartis Investigative Site, Poprad, Slovakia
  - Novartis Investigative Site, Ružomberok, Slovakia
  - Novartis Investigative Site, Bratislava
- Thailand (3):
  - Novartis Investigative Site, Muang, Thailand
  - Novartis Investigative Site, Rajathevee, Thailand
  - Novartis Investigative Site, Ratchathewi, Thailand
- Turkey (Türkiye) (6):
  - Novartis Investigative Site, Adana, Turkey
  - Novartis Investigative Site, Bursa, Turkey
  - Novartis Investigative Site, Gaziantep, Turkey
  - Novartis Investigative Site, Istanbul, Turkey
  - Novartis Investigative Site, Izmir, Turkey
  - Novartis Investigative Site, Talas / Kayseri
- Ukraine (5):
  - Novartis Investigative Site, Dnipropetrovsk, Ukraine
  - Novartis Investigative Site, Donetsk, Ukraine
  - Novartis Investigative Site, Kharkiv, Ukraine
  - Novartis Investigative Site, Kyiv, Ukraine
  - Novartis Investigative Site, Vinnytsia, Ukraine

RESULTS

PARTICIPANT FLOW:
Groups:
- Mometasone Furoate 80 ug Daily Via the Concept1 Device: Mometasone furoate (MF) delivered via Concept1, 80 μg daily in the evening
- Mometasone Furoate 200 ug Daily Via the Twisthaler® Device: Mometasone furoate delivered via Twisthaler®, 200 μg daily in the evening
- Mometasone Furoate 320 ug Daily Via the Concept1 Device: Mometasone furoate (MF) delivered via Concept1, 320 μg daily in the evening
- Mometasone Furoate 800 ug Via the Twisthaler® Device: Mometasone furoate delivered via Twisthaler®, 800 μg daily in the evening
Period: Overall Study
Arm/Group | Mometasone Furoate 80 ug Daily Via the Concept1 Device | Mometasone Furoate 200 ug Daily Via the Twisthaler® Device | Mometasone Furoate 320 ug Daily Via the Concept1 Device | Mometasone Furoate 800 ug Via the Twisthaler® Device
Started | 188 | 181 | 184 | 186
Safety Set (SAF) | 186 | 180 | 183 | 186
Completed | 175 | 173 | 178 | 176
Not Completed | 13 | 8 | 6 | 10
Not completed — Withdrawal by Subject | 6 | 2 | 0 | 2
Not completed — Administrative | 3 | 1 | 2 | 0
Not completed — Protocol Violation | 3 | 3 | 3 | 5
Not completed — Adverse Event | 1 | 2 | 1 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mometasone Furoate 80 ug Daily Via the Concept1 Device | Mometasone Furoate 200 ug Daily Via the Twisthaler® Device | Mometasone Furoate 320 ug Daily Via the Concept1 Device | Mometasone Furoate 800 ug Via the Twisthaler® Device | Total
Number analyzed (Participants) | 188 | 181 | 184 | 186 | 739
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.4 (16.33) | 45.9 (15.56) | 46.0 (16.18) | 45.5 (16.57) | 45.4 (16.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 94 | 113 | 97 | 402
  Male | 90 | 87 | 71 | 89 | 337

OUTCOME MEASURES:

1. Primary Outcome: Trough Forced Expiratory Volume in 1 Second (FEV1)
Description: Forced Expiratory Volume in 1 second (FEV1) was measured via spirometry conducted according to internationally accepted standards. Measurements were taken on day 29 after treatment.
Time Frame: Day 29
Population: The Full Analysis Set (FAS) includes all randomized subjects who received at least one dose of study drug with available data for analysis.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Mometasone Furoate 80 ug Daily Via the Concept1 Device | Mometasone Furoate 200 ug Daily Via the Twisthaler® Device | Mometasone Furoate 320 ug Daily Via the Concept1 Device | Mometasone Furoate 800 ug Via the Twisthaler® Device
Number analyzed (Participants) | 171 | 165 | 172 | 173
Liters | 2.139 (0.0281) | 2.071 (0.0283) | 2.187 (0.0281) | 2.162 (0.0279)

2. Secondary Outcome: Trough Forced Expiratory Volume in 1 Second (FEV1) After Days 8, 15 and 22 of Treatment
Description: Forced Expiratory Volume in 1 second (FEV1) was measured via spirometry conducted according to internationally accepted standards. Measurements were taken on days 8, 15 and 22 after treatment. Data within 6 hr of rescue medication use is excluded from this analysis.
Time Frame: Days 8, 15 and 22
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Mometasone Furoate 80 ug Daily Via the Concept1 Device | Mometasone Furoate 200 ug Daily Via the Twisthaler® Device | Mometasone Furoate 320 ug Daily Via the Concept1 Device | Mometasone Furoate 800 ug Via the Twisthaler® Device
Number analyzed (Participants) | 179 | 173 | 181 | 181
Liters
  Day 8 (n=178,173,181,181) | 2.069 (0.0252) | 2.057 (0.0253) | 2.113 (0.0251) | 2.111 (0.0250)
  Day 15 (n=179,171,177,178) | 2.095 (0.0254) | 2.048 (0.0258) | 2.134 (0.0257) | 2.135 (0.0255)
  Day 22 (n=174,170,177,177) | 2.126 (0.0284) | 2.071 (0.0286) | 2.175 (0.0283) | 2.146 (0.0282)

3. Secondary Outcome: Forced Vital Capacity (FVC) at All Time Points
Description: Forced Vital Capacity (FVC) is the amount of air which can be forcibly exhaled from the lungs after taking the deepest breath possible. Data within 6 hr of rescue medication use is excluded from this analysis. Mixed model: FVC = treatment + gender+ baseline FVC + age + level of asthma control + region + center (region) + error. Center is included as a random effect nested within region.
Time Frame: Days 1, 8, 15, 22, 28 and 29 at all time points
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Mometasone Furoate 80 ug Daily Via the Concept1 Device | Mometasone Furoate 200 ug Daily Via the Twisthaler® Device | Mometasone Furoate 320 ug Daily Via the Concept1 Device | Mometasone Furoate 800 ug Via the Twisthaler® Device
Number analyzed (Participants) | 178 | 172 | 179 | 174
Liters
  Day 1/30 min post-dose (n=172,172,175,173) | 2.892 (0.0208) | 2.893 (0.0207) | 2.861 (0.0209) | 2.897 (0.0208)
  Day 1/1 hr post-dose (n=178,169,174,175) | 2.930 (0.0234) | 2.913 (0.0238) | 2.943 (0.0238) | 2.946 (0.0235)
  Day 8/50 min pre-dose (n=174,171,179,174) | 3.111 (0.0325) | 3.096 (0.0325) | 3.134 (0.0321) | 3.139 (0.0324)
  Day 8/15 min pre-dose (n=176,172,179,174) | 3.099 (0.0324) | 3.074 (0.0324) | 3.121 (0.0321) | 3.125 (0.0323)
  Day 15 /50 min pre-dose (n=175,169,170,169) | 3.134 (0.0342) | 3.090 (0.0347) | 3.168 (0.0348) | 3.155 (0.0348)
  Day 15/15 min pre-dose (n=176,168,176,167) | 3.109 (0.0343) | 3.076 (0.0348) | 3.137 (0.0345) | 3.127 (0.0348)
  Day 22/50 min pre-dose (n=172,167,174,169) | 3.136 (0.0356) | 3.091 (0.0359) | 3.203 (0.0355) | 3.152 (0.0357)
  Day 22/15 min pre-dose (n=169,170,174,172) | 3.134 (0.0365) | 3.096 (0.0363) | 3.198 (0.0362) | 3.157 (0.0361)
  Day 28/50 min pre-dose (n=172,168,176,172) | 3.146 (0.0342) | 3.115 (0.0345) | 3.184 (0.0340) | 3.180 (0.0342)
  Day 28/15 min pre-dose (n=170,165,174, 170) | 3.135 (0.0345) | 3.095 (0.0348) | 3.153 (0.0343) | 3.161 (0.0344)
  Day 28/30 min post-dose (n=175,166,174,170) | 3.132 (0.0341) | 3.092 (0.0346) | 3.151 (0.0343) | 3.184 (0.0343)
  Day 28/30 min post-dose (n=173,167,172,172) | 3.140 (0.0351) | 3.084 (0.0353) | 3.158 (0.0353) | 3.161 (0.0350)
  Day 29/23hr 10 min post-dose (n=173,162,172,168) | 3.160 (0.0342) | 3.113 (0.0348) | 3.216 (0.0343) | 3.194 (0.0344)
  Day 29/23hr 45 min post-dose (n=172,161, 175,170) | 3.165 (0.0355) | 3.090 (0.0363) | 3.192 (0.0353) | 3.158 (0.0355)

4. Secondary Outcome: Forced Expiratory Flow Between 25% and 75% (FEF25-75%) at All Time Points
Description: The Forced Expiratory Flow (FEF) 25%-75% measurement describes the amount of air expelled from the lungs during the middle half (25% - 75%) of the forced vital capacity test and is measured using spirometry.
Time Frame: Days 1, 8, 15, 22, 28 and 29 at all time points
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters per second
Arm/Group | Mometasone Furoate 80 ug Daily Via the Concept1 Device | Mometasone Furoate 200 ug Daily Via the Twisthaler® Device | Mometasone Furoate 320 ug Daily Via the Concept1 Device | Mometasone Furoate 800 ug Via the Twisthaler® Device
Number analyzed (Participants) | 178 | 172 | 179 | 174
Liters per second
  Day 1/30 min post-dose (n=172,172,175,172) | 1.308 (0.0181) | 1.300 (0.0182) | 1.309 (0.0182) | 1.308 (0.0182)
  Day 1/1 hr post-dose (n=178,169,174,174) | 1.337 (0.0197) | 1.327 (0.0201) | 1.316 (0.0201) | 1.345 (0.0199)
  Day 8/50 min pre-dose (n=173,171,179,174) | 1.457 (0.0323) | 1.449 (0.0322) | 1.519 (0.0317) | 1.525 (0.0321)
  Day 8/15 min pre-dose (n=175,172,179,173) | 1.458 (0.0329) | 1.466 (0.0328) | 1.542 (0.0325) | 1.566 (0.0328)
  Day 15 /50 min pre-dose (n=175,169,170,169) | 1.509 (0.0317) | 1.430 (0.0321) | 1.514 (0.0320) | 1.544 (0.0321)
  Day 15/15 min pre-dose (n=175,168,176,167) | 1.494 (0.0322) | 1.414 (0.0326) | 1.520 (0.0321) | 1.561 (0.0327)
  Day 22/50 min pre-dose (n=171,167,174,169) | 1.511 (0.0350) | 1.440 (0.0353) | 1.565 (0.0348) | 1.555 (0.0351)
  Day 22/15 min pre-dose (n=168,170,174,172) | 1.540 (0.0365) | 1.476 (0.0362) | 1.600 (0.0361) | 1.591 (0.0361)
  Day 28/50 min pre-dose (n=171,168,176,172) | 1.504 (0.0353) | 1.458 (0.0354) | 1.581 (0.0350) | 1.598 (0.0351)
  Day 28/15 min pre-dose (n=169,165,174, 170) | 1.529 (0.0357) | 1.481 (0.0359) | 1.574 (0.0354) | 1.584 (0.0355)
  Day 28/30 min post-dose (n=175,166,174,170) | 1.558 (0.0362) | 1.457 (0.0368) | 1.557 (0.0364) | 1.615 (0.0364)
  Day 28/30 min post-dose (n=172,167,172,172) | 1.566 (0.0367) | 1.460 (0.0369) | 1.577 (0.0368) | 1.593 (0.0365)
  Day 29/23hr 10 min post-dose (n=172,162,172,168) | 1.537 (0.0369) | 1.451 (0.0376) | 1.604 (0.0369) | 1.584 (0.0371)
  Day 29/23hr 45 min post-dose (n=171,161, 175,170) | 1.550 (0.0370) | 1.438 (0.0378) | 1.576 (0.0366) | 1.571 (0.0369)

5. Secondary Outcome: Forced Expiratory Volume in 1 Second Forced Vital Capacity (FEV1/FVC) Percent at All Time Points
Description: Forced Expiratory Volume in 1 second (FEV1)/Forced Vital Capacity (FVC) was measured via spirometry conducted according to internationally accepted standards. Data within 6 hr of rescue medication use is excluded from this analysis.
Time Frame: Days 1, 8, 15, 22, 28 and 29 at all time points
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent
Arm/Group | Mometasone Furoate 80 ug Daily Via the Concept1 Device | Mometasone Furoate 200 ug Daily Via the Twisthaler® Device | Mometasone Furoate 320 ug Daily Via the Concept1 Device | Mometasone Furoate 800 ug Via the Twisthaler® Device
Number analyzed (Participants) | 178 | 172 | 179 | 175
Percent
  Day 1/30 min post-dose (n=172,172,175,173) | 65.043 (0.2548) | 64.898 (0.2556) | 65.184 (0.2559) | 64.898 (0.2554)
  Day 1/1 hr post-dose (n=178,169,174,175) | 65.177 (0.2833) | 64.833 (0.2890) | 65.005 (0.2885) | 65.072 (0.2845)
  Day 8/50 min pre-dose (n=174,171,179,175) | 66.566 (0.4281) | 66.301 (0.4286) | 67.344 (0.4222) | 66.568 (0.4264)
  Day 8/15 min pre-dose (n=176,172,179,174) | 66.595 (0.4259) | 66.790 (0.4262) | 67.778 (0.4224) | 67.156 (0.4252)
  Day 15 /50 min pre-dose (n=176,169,170,169) | 67.007 (0.4329) | 66.122 (0.4398) | 67.487 (0.4395) | 67.139 (0.4407)
  Day 15/15 min pre-dose (n=176,168,176,167) | 66.878 (0.4370) | 66.006 (0.4443) | 67.607 (0.4384) | 67.514 (0.4456)
  Day 22/50 min pre-dose (n=172,167,174,169) | 67.081 (0.4594) | 66.567 (0.4643) | 67.831 (0.4584) | 67.742 (0.4615)
  Day 22/15 min pre-dose (n=169,170,174,172) | 67.403 (0.4657) | 66.885 (0.4629) | 68.143 (0.4622) | 67.895 (0.4612)
  Day 28/50 min pre-dose (n=172,168,176,172) | 67.128 (0.4584) | 66.835 (0.4615) | 68.124 (0.4567) | 67.810 (0.4578)
  Day 28/15 min pre-dose (n=170,165,174, 170) | 67.503 (0.4813) | 67.296 (0.4854) | 68.255 (0.4796) | 67.878 (0.4804)
  Day 28/30 min post-dose (n=175,166,174,170) | 67.700 (0.4723) | 67.013 (0.4796) | 68.031 (0.4755) | 68.126 (0.4755)
  Day 28/30 min post-dose (n=173,167,172,172) | 67.945 (0.4703) | 66.832 (0.4741) | 68.243 (0.4736) | 68.057 (0.4698)
  Day 29/23hr 10 min post-dose (n=173,162,172,168) | 67.427 (0.4639) | 66.711 (0.4736) | 68.265 (0.4654) | 67.592 (0.4676)
  Day 29/23hr 45 min post-dose (n=172,161, 175,170) | 67.630 (0.4694) | 66.541 (0.4806) | 67.961 (0.4667) | 67.831 (0.4692)

6. Secondary Outcome: Change From Baseline in Mean Morning and Evening Peak Expiratory Flow Rate (PEFR) Over 4 Weeks of Treatment
Description: Peak expiratory flow rate (PEFR) was measured via electronice Peak flow meter by patient at home. Mixed model used: change from baseline in the mean evening PEFR = treatment + age + gender + baseline evening PEFR + level of asthma control + region + center (region)+ error. Center is included as a random effect nested within region.
Time Frame: Baseline and week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters per min
Arm/Group | Mometasone Furoate 80 ug Daily Via the Concept1 Device | Mometasone Furoate 200 ug Daily Via the Twisthaler® Device | Mometasone Furoate 320 ug Daily Via the Concept1 Device | Mometasone Furoate 800 ug Via the Twisthaler® Device
Number analyzed (Participants) | 177 | 172 | 175 | 182
Liters per min
  Morning 4 wks-baseline (n=177,171, 175, 182) | -4.952 (4.1929) | 3.955 (4.2616) | 2.785 (4.2349) | 1.606 (4.1464)
  Evening 4 wks-baseline (n=176, 172, 174, 179) | 1.354 (3.9003) | 0.293 (3.9477) | -0.644 (3.9427) | 6.287 (3.8826)

7. Secondary Outcome: Change From Baseline in Asthma Control Questionnaire (ACQ-5) by Visit
Description: Asthma symptoms were evaluated by the Asthma Control Questionnaire (ACQ). The ACQ-5 has five questions of the asthma symptoms to be answered by the patient. The overall score is the average of the 5 questions; a minimum overall score of 0 = good control of asthma whereas a maximum overall score of 6 = poor control of asthma. A negative change in score indicates improvement in symptoms. MIXED model: Change from baseline in ACQ-5 = treatment + gender + baseline ACQ-5 score + age + level of asthma control + region + center (region) + error. Center is included as a random effect nested within region. - Baseline ACQ-5 is defined as the questionnaire completed on Day 1 (randomization).
Time Frame: Baseline, days 8,15,22 and 29
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Mometasone Furoate 80 ug Daily Via the Concept1 Device | Mometasone Furoate 200 ug Daily Via the Twisthaler® Device | Mometasone Furoate 320 ug Daily Via the Concept1 Device | Mometasone Furoate 800 ug Via the Twisthaler® Device
Number analyzed (Participants) | 180 | 176 | 182 | 182
Units on a scale
  Day 8-baseline (n=179,176,182,182) | -0.662 (0.0543) | -0.730 (0.0546) | -0.908 (0.0540) | -0.890 (0.0538)
  Day 15-baseline(n=180,174,179,178) | -0.899 (0.0590) | -0.908 (0.0599) | -1.117 (0.0595) | -0.973 (0.0593)
  Day 22-baseline (n=178,173,178,177) | -0.994 (0.0620) | -0.982 (0.0628) | -1.262 (0.0622) | -1.097 (0.0622)
  Day 29-baseline (n=179,176,181,182) | -1.079 (0.0630) | -1.109 (0.602) | -1.329 (0.0632) | -1.162 (0.0625)

8. Secondary Outcome: Change From Baseline in Mean Daily Number of Puffs of Rescue Medication Over 4 Weeks of Treatment
Description: Rescue medication data recorded during the 14 day run-in period is used to calculate the baseline. - Total number of puffs of rescue medication per day over the full 4 weeks is calculated and divided by the total number of days with non-missing rescue medication data to derive the mean daily number of puffs of rescue medication taken for the subject. - MIXED model: Change = treatment + gender + baseline mean daily number of puffs + age + level of asthma control + region + center (region) + error. Center is included as a random effect nested within region.
Time Frame: Baseline and 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: number of puffs
Arm/Group | Mometasone Furoate 80 ug Daily Via the Concept1 Device | Mometasone Furoate 200 ug Daily Via the Twisthaler® Device | Mometasone Furoate 320 ug Daily Via the Concept1 Device | Mometasone Furoate 800 ug Via the Twisthaler® Device
Number analyzed (Participants) | 177 | 172 | 175 | 181
number of puffs | -0.456 (0.0972) | -0.391 (0.0985) | -0.600 (0.0981) | -0.677 (0.0963)

9. Secondary Outcome: Percentage of Days With no Rescue Medication Use Over 4 Weeks of Treatment
Description: Mixed model used: percentage of days with no rescue medication use = treatment + age + gender + baseline percentage of days with no rescue use + level of asthma control + region + center (region) + error. Center is included as a random effect nested within region.
  A day with no rescue use is defined from diary data as any day where the subject does not use any puffs of rescue medication.
  The total number of days with no rescue use over the 4 week treatment period is divided by the total number of evaluable days in order to derive the percentage of days with no rescue use.
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage days
Arm/Group | Mometasone Furoate 80 ug Daily Via the Concept1 Device | Mometasone Furoate 200 ug Daily Via the Twisthaler® Device | Mometasone Furoate 320 ug Daily Via the Concept1 Device | Mometasone Furoate 800 ug Via the Twisthaler® Device
Number analyzed (Participants) | 124 | 116 | 117 | 113
percentage days | 74.148 (2.2576) | 75.236 (2.3291) | 75.157 (2.3044) | 80.578 (2.3476)

10. Secondary Outcome: Fractional Exhaled Nitric Oxide (FeNO)
Description: FeNO is widely accepted as a non-invasive marker for airway inflammation such as asthma and conducted according to published guideline. FeNO was measured on days 15 and 29 after treatment.
Time Frame: Days 15 and 29
Population: as for outcome 1
Measure: Mean (Standard Error); unit: ppm
Arm/Group | Mometasone Furoate 80 ug Daily Via the Concept1 Device | Mometasone Furoate 200 ug Daily Via the Twisthaler® Device | Mometasone Furoate 320 ug Daily Via the Concept1 Device | Mometasone Furoate 800 ug Via the Twisthaler® Device
Number analyzed (Participants) | 142 | 143 | 145 | 150
ppm
  Day 15 (n= 142, 139, 139, 149) | 25.286 (1.2983) | 26.762 (1.3201) | 19.098 (1.3246) | 21.017 (1.2911)
  Day 29 (n=141, 143, 145, 150) | 23.777 (1.3078) | 27.055 (1.3035) | 18.468 (1.2952) | 19.981 (1.2803)

11. Secondary Outcome: Plasma Cortisol Concentrations
Description: Blood samples were taken from each subject participating in the study post dose at day 1 and week 4. Cortisol concentrations were evaluated. Results are presented as nmol/L
Time Frame: Baseline, days 1 and 28
Population: The safety set includes all subjects who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Mometasone Furoate 80 ug Daily Via the Concept1 Device | Mometasone Furoate 200 ug Daily Via the Twisthaler® Device | Mometasone Furoate 320 ug Daily Via the Concept1 Device | Mometasone Furoate 800 ug Via the Twisthaler® Device
Number analyzed (Participants) | 183 | 178 | 179 | 181
nmol/L
  Baseline (n= 183, 178, 179, 181) | 150.040 (80.3928) | 143.132 (88.4206) | 143.791 (85.8696) | 150.108 (88.6815)
  Day 1/1 Hr (n=179, 177,174, 176) | 118.130 (92.7539) | 106.965 (81.5160) | 107.526 (74.3770) | 115.489 (79.3869)
  Day 28/-25 Mins (n= 172, 169, 174, 172) | 140.760 (73.3567) | 140.604 (72.8885) | 143.555 (82.4961) | 145.484 (92.2940)
  Day 28/1 Hr (n= 172, 168, 174, 170) | 105.399 (68.9416) | 107.931 (70.7374) | 105.468 (57.9029) | 110.477 (77.2220)

ADVERSE EVENTS:
Groups:
- Total: Total
Arm/Group | Mometasone Furoate 80 ug Daily Via the Concept1 Device | Mometasone Furoate 200 ug Daily Via the Twisthaler® Device | Mometasone Furoate 320 ug Daily Via the Concept1 Device | Mometasone Furoate 800 ug Via the Twisthaler® Device | Total
Serious Adverse Events (participants affected / at risk) | 0/186 | 0/180 | 1/183 | 0/186 | 1/735
Other Adverse Events (participants affected / at risk) | 13/186 | 17/180 | 15/183 | 8/186 | 53/735
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mometasone Furoate 80 ug Daily Via the Concept1 Device (N=186) | Mometasone Furoate 200 ug Daily Via the Twisthaler® Device (N=180) | Mometasone Furoate 320 ug Daily Via the Concept1 Device (N=183) | Mometasone Furoate 800 ug Via the Twisthaler® Device (N=186) | Total (N=735)
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mometasone Furoate 80 ug Daily Via the Concept1 Device (N=186) | Mometasone Furoate 200 ug Daily Via the Twisthaler® Device (N=180) | Mometasone Furoate 320 ug Daily Via the Concept1 Device (N=183) | Mometasone Furoate 800 ug Via the Twisthaler® Device (N=186) | Total (N=735)
Nasopharyngitis (Infections and infestations) | 3 | 7 | 6 | 2 | 18
Blood cortisol decreased (Investigations) | 4 | 3 | 5 | 6 | 18
Headache (Nervous system disorders) | 6 | 5 | 5 | 0 | 16
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 1 | 0 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.